CLINICAL TRIAL: NCT03992482
Title: A Phase I/II Randomized, Placebo-controlled, Double-Blind, Single-Center, Tolerability and Preliminary Efficacy Clinical Trial of Intravenous Immunoglobulin (IVIG) Eye Drops in Patients With Dry Eye Disease
Brief Title: IVIG-eye Drops Treatment for Dry Eye Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sandeep Jain, MD (Other)
Responsible Party: Sponsor-Investigator, Sandeep Jain, MD, Professor, University of Illinois at Chicago
Organization: University of Illinois at Chicago (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-0263
Record Dates: First submitted 2019-06-13; First posted 2019-06-20 (Actual); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Dry Eye
Keywords: Dry Eye; Intravenous Immunoglobulin (IVIG) Eye Drops; Treatment; ocular Graft-vs-Host Disease (oGVHD)
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IVIG-Eye Drop (Experimental): Intravenous Immunoglobulin (IVIG), 4 mg/ml (0.4%) eye drops two times a day for eight weeks
  Interventions: Drug: Intravenous Immune Globulin (IVIG)
- Placebo-Eye Drop (Placebo Comparator): Normal Saline Eye Drops (0.9% NaCl)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intravenous Immune Globulin (IVIG) — Intravenous Immunoglobulin (IVIG), 4 mg/ml (0.4%) eye drops two times a day for eight weeks
  Arms: IVIG-Eye Drop
Drug: Placebo — Normal Saline Eye Drops (0.9% NaCl) two times a day for eight weeks
  Arms: Placebo-Eye Drop

SUMMARY:
The main objective of this study is to establish whether patients with Dry Eye Disease are able to safely tolerate receiving Intravenous Immunoglobulin (IVIG) eye drops two times a day for eight weeks (primary 'safety and tolerability' objective). The exploratory objective is to investigate the preliminary efficacy of the use of IVIG eye drops in treating Dry Eye Disease (exploratory efficacy objective) to estimate the effectiveness of the trial intervention and collecting data to inform the design of a future definitive trial.

This will be a Randomized controlled trial, in which a total of 28 subjects will be enrolled at 1 clinical site. Subjects will be randomly assigned to one of two groups (#1, #2), with 14 subjects per group. One group will be given placebo (Normal saline eye drops) and the other group will be given eye drops containing the study drug (IVIG).

ELIGIBILITY:
Inclusion Criteria:

1. Sign and date the informed consent form approved by the Institutional Review Board (IRB)
2. ≥ 18 years of age
3. Demonstrate at least any 2 of the following signs in the same eye or a sign and symptom.

   1. Conjunctival staining present ≥ 1 (out of possible score of 6 per eye)
   2. Corneal staining present ≥ 2 (out of a possible score of 15 per eye)
   3. Tear film break up time (TFBUT) ≤ 7 seconds
   4. Schirmer's test ≥ 0 to ≤ 9 mm/5min
   5. Superior Limbic Keratoconjunctivitis (SLK) pattern staining ≥ 1
   6. Meiboscale grade ≥ 2
   7. Validated Bulbar Redness ≥ 40
   8. Demonstrate symptoms of dry eye disease Ocular Surface Disease Index (OSDI) score of at least ≥ 13.
   9. Demonstrate Symptom Intensity Assessment of ≥ 3.
4. Patient reported dry eye-related ocular symptoms for at least 6 months before the Screening Visit and use or desire to use artificial tears on average 2 times per day in the 2 weeks preceding the screening visit
5. Intraocular pressure (IOP) ≥ 5 mmHg and ≤ 22 mmHg in each eye
6. Women of child-bearing potential must agree to use a reliable method of contraception during study participation and must demonstrate a negative pregnancy test at the Screening Visit
7. Be willing/able to return for all study visits and to follow instructions from the study investigator and his/her staff
8. Ocular Surface Wash Anti-Citrullinated Protein Antibody (ACPA) value of > 4.4 units in either eye at any time in the past.

Exclusion Criteria:

1. Allergic to IVIG or any similar products, or excipients of IVIG eye drops 4 mg/ml.
2. Use of contact lenses within the last 2-weeks prior to the baseline Visit.
3. Use of Allogenic serum or plasma eye drops within the last 2-weeks prior to the baseline Visit.
4. Unwilling to commit to no use of contact lenses for the duration of the study.
5. Pregnant or nursing/lactating
6. Participation in a study of an investigational drug or device within the 30 days preceding the Screening Visit
7. Current diagnosis of any of the following ocular conditions:

   i) Acute allergic conjunctivitis ii) Active infection (e.g. bacterial, viral, protozoan or fungal infection of the cornea, conjunctiva, lacrimal gland, lacrimal sac or eyelids) iii) Active intraocular inflammation (e.g., retinitis, choroiditis, uveitis)
8. A cognitive or psychiatric deficit that precludes informed consent or ability to perform
9. Vulnerable populations, such as neonates, pregnant women, children, prisoners, institutionalized individuals, or others who may be considered vulnerable populations.
10. Have active drug/alcohol dependence or abuse.
11. The corneal epithelial defect is larger than 1 mm2 in either eye.
12. Active ocular infection or ocular allergies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Jain, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Illinois Eye and Ear Infirmary, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin-Nares E, Hernandez-Molina G. Novel autoantibodies in Sjogren's syndrome: A comprehensive review. Autoimmun Rev. 2019 Feb;18(2):192-198. doi: 10.1016/j.autrev.2018.09.003. Epub 2018 Dec 18. PMID 30572138
- [Background] Dourmishev LA, Guleva DV, Miteva LG. Intravenous Immunoglobulins: Mode of Action and Indications in Autoimmune and Inflammatory Dermatoses. Int J Inflam. 2016;2016:3523057. doi: 10.1155/2016/3523057. Epub 2016 Jan 18. PMID 26885437
- [Background] Mun C, Gulati S, Tibrewal S, Chen YF, An S, Surenkhuu B, Raju I, Buwick M, Ahn A, Kwon JE, Atassi N, Pradeep A, Rondelli D, Jain S. A Phase I/II Placebo-Controlled Randomized Pilot Clinical Trial of Recombinant Deoxyribonuclease (DNase) Eye Drops Use in Patients With Dry Eye Disease. Transl Vis Sci Technol. 2019 May 2;8(3):10. doi: 10.1167/tvst.8.3.10. eCollection 2019 May. PMID 31110911
- [Background] An S, Raju I, Surenkhuu B, Kwon JE, Gulati S, Karaman M, Pradeep A, Sinha S, Mun C, Jain S. Neutrophil extracellular traps (NETs) contribute to pathological changes of ocular graft-vs.-host disease (oGVHD) dry eye: Implications for novel biomarkers and therapeutic strategies. Ocul Surf. 2019 Jul;17(3):589-614. doi: 10.1016/j.jtos.2019.03.010. Epub 2019 Apr 6. PMID 30965123
- See also: Related Info — http://chicago.medicine.uic.edu/directory/name/sandeep-jain-md-jain/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the clinical practice of the investigator at the time of their routine eye examination visit. The clinical practice is located in the Illinois Eye and Ear Infirmary (EEI), the University of Illinois at Chicago (UIC). The first participant was enrolled on 6 May 2019, and the last participant was enrolled on 7 June 2019.
Period: Overall Study
Arm/Group | IVIG-Eye Drop | Placebo-Eye Drop
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVIG-Eye Drop | Placebo-Eye Drop | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [47 to 66] | 65 [51.2 to 71] | 62 [48.5 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 8 | 11 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27
Diagnosis [Count of Participants; unit: Participants]
  Auto-immune tear deficient DED | 7 | 6 | 13
  ocular GVHD | 6 | 1 | 7
  Non-autoimmune tear deficient DED | 0 | 5 | 5
  Meibomian Gland Dysfunction (MGD) | 0 | 2 | 2
OSDI [Median (Inter-Quartile Range); unit: units on a scale] — Ocular Surface Disease Index (OSDI), 12-item questionnaire, assesses symptom of ocular irritation in dry eye disease (DED) and how it affects functioning related to vision in past week. It has 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients rate their responses on 0 to 4 scale with 0 being "none of the time" and 4 being "all of the time." OSDI score range from 0-100 with score 0-12 being normal, 13-22 being mild DED, 23-32 being moderate DED, and >33 being severe DED. OSDI=[(sum of scores for questions answered)×100]/[(total questions answered)×4]
  units on a scale | 52.3 [35 to 58.3] | 40.9 [35 to 59.4] | 43.18 [35 to 58.8]
Corneal Staining [Median (Inter-Quartile Range); unit: units on a scale] — Corneal staining score as measured by Lissamine Green dye staining using National Eye Institute (NEI) grading scale. Dye was applied to each eye and a slit lamp was used to observe corneal staining. NEI scale relies on a chart that divides the cornea into 5 sections and assigns a value from 0 (absent) to 3 (severe) to each section, based on the density of punctate staining, final staining score being the sum of individual section scores with a range of 0 (minimum) -15 (maximum) points. Complete corneal staining clearance with Lissamine dye defined as a score of 0 indicating the best outcome.
  units on a scale | 5 [2.25 to 7.75] | 2 [1 to 4.25] | 3 [2 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Tolerability: The Primary Tolerability Endpoint is the Test Substance Tolerance (Visual Analog Scale) at 8 Weeks (56 Days)
Description: Subjects will assess their tolerance to the administration of the test medication (placebo/ study drug), utilizing a Visual Analog Scale (VAS). The VAS is a 100 mm horizontal line with verbal descriptors at either end. Subjects will place a single slash mark across the horizontal line between the end labeled "completely intolerable" (0 mm) and "easily tolerable" (100mm). The VAS ratings will be completed after administration of the test medication on Day 1 (post-dose), week 4 and week 8.
Time Frame: 8 Weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IVIG-Eye Drop | Placebo-Eye Drop
Number analyzed (Participants) | 13 | 14
score on a scale | 100 [100 to 100] | 100 [100 to 100]
Statistical Analysis 1: Comparison: IVIG-Eye Drop vs Placebo-Eye Drop; Test type: Other; p = 1.000, Kruskal-Wallis

2. Other Pre Specified Outcome: The Change in the Ocular Surface Disease Index (OSDI) Which is a Patient's Subjective Rating Scale
Description: Ocular Surface Disease Index (OSDI), a 12-item questionnaire, assesses symptom of ocular irritation in dry eye disease (DED) and how it affects functioning related to vision in the past week. It has 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients rate their responses on 0 to 4 scale with 0 being "none of the time" and 4 being "all of the time." OSDI score range from 0-100 with score 0-12 being normal, 13-22 being mild DED, 23-32 being moderate DED, and >33 being severe DED. OSDI=[(sum of scores for questions answered)×100]/[(total questions answered)×4]
Time Frame: Between baseline and at 8 weeks of treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IVIG-Eye Drop | Placebo-Eye Drop
Number analyzed (Participants) | 13 | 14
score on a scale | -20.9 [-24.43 to -15.00] | 0.00 [-12.08 to 4.28]
Statistical Analysis 1: Comparison: IVIG-Eye Drop vs Placebo-Eye Drop; Test type: Other; p = 0.0044, Mixed Models Analysis

3. Other Pre Specified Outcome: Change in Corneal Staining Score as Measured by Lissamine Dye Staining
Description: Corneal staining score as measured by Lissamine Green dye staining using National Eye Institute (NEI) grading scale. Dye was applied to each eye and a slit lamp was used to observe corneal staining. NEI scale relies on a chart that divides the cornea into 5 sections and assigns a value from 0 (absent) to 3 (severe) to each section, based on the density of punctate staining, final staining score being the sum of individual section scores with a range of 0 (minimum) -15 (maximum) points. Complete corneal staining clearance with Lissamine dye defined as a score of 0 indicating the best outcome.
Time Frame: Between baseline and at 8 weeks of treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Units Other Than Participants: Eye
Arm/Group | IVIG-Eye Drop | Placebo-Eye Drop
Number analyzed (Participants) | 13 | 14
Number analyzed (Eye) | 26 | 28
score on a scale | -1.50 [-3.50 to 0.00] | 0.00 [0.00 to 1.25]
Statistical Analysis 1: Comparison: IVIG-Eye Drop vs Placebo-Eye Drop; Test type: Other; p = 0.0002, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Between baseline and 8-weeks of treatment
Arm/Group | IVIG-Eye Drop | Placebo-Eye Drop
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 5/13 | 8/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IVIG-Eye Drop (N=13) | Placebo-Eye Drop (N=14)
Ocular discomfort (Eye disorders) | 2 | 5
Pain (Eye disorders) | 0 | 1
Tearing (Eye disorders) | 0 | 2
Blurring of vision (Eye disorders) | 2 | 4
Light sensitivity (Eye disorders) | 1 | 5
Dryness (Eye disorders) | 2 | 4
Redness (Eye disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Outcomes of this clinical trial shouldn't be over-interpreted for benefit. Accurate assessment of therapeutic implications of IVIG eye drops will only be possible after adequately powered definitive pivotal trials. Small sample size is a limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT03992482/Prot_SAP_000.pdf